CLINICAL TRIAL: NCT05462743
Title: Artificial Intelligence-assisted Confocal Laser Endomicroscopy Identification of Intestinal Metaplasia Severity for Gastric Cancer Risk Assessment
Brief Title: Artificial Intelligence-assisted Confocal Laser Endomicroscopy Identification of Intestinal Metaplasia Severity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Other Study IDs: 2022-SDU-QILU-122
Record Dates: First submitted 2022-07-09; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Intestinal Metaplasia; Artificial Intelligence; Confocal Laser Endomicroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — When a gastric mucosal leison is found using white light endoscopy, endoscopist will observe this lesion using pCLE and then take biopsy for histology examination.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group for training the algorithm: This group of images is used for training the algorithm of the artifical intelligence
- group for testing the algorithm: This group of images is used for testing the algorithm of the artifical intelligence

SUMMARY:
Currently, the Correa cascade is a widely accepted model of gastric carcinogenesis. Intestinal metaplasia is a high risk factor for gastric cancer. According to Sydney criteria, mild intestinal metaplasia was not associated with gastric cancer, while moderate to severe intestinal metaplasia was strongly associated with the development of gastric cancer. Because intestinal metaplasia is distributed in various forms, the use of white light endoscopy lacks specificity, and the consistency with histopathological diagnosis is poor; Pathological biopsy is still needed to make a diagnosis. At present, national guidelines suggest that OLGIM score should be used to evaluate the risk of gastric cancer, and patients with OLGIM grade III/IV should be monitored by close gastroscopy. However, it requires at least four biopsies, which is clinically infeasible. Confocal laser endomicroscopy allows real-time observation of living tissue, comparable to pathological findings.

DETAILED DESCRIPTION:
Gastric cancer is a common malignant tumor in digestive system diseases. Currently, the Correa cascade is a widely accepted model of gastric carcinogenesis. Intestinal metaplasia is a high risk factor for gastric cancer and is considered a precancerous condition of intestinal type gastric cancer. According to Sydney criteria, mild intestinal metaplasia was not associated with gastric cancer, while moderate to severe intestinal metaplasia was strongly associated with the development of gastric cancer. Because intestinal metaplasia is distributed in various forms, the use of white light endoscopy lacks specificity, and the consistency with histopathological diagnosis is poor; Pathological biopsy is still needed to make a diagnosis. At present, our national guidelines suggest that OLGIM score should be used to evaluate the risk of gastric cancer, and patients with OLGIM grade III/IV should be monitored by close gastroscopy. However, it requires at least four biopsies, which is clinically infeasible. Confocal laser endomicroscopy allows real-time observation of living tissue, comparable to pathological findings. Therefore, we established artificial intelligence-assisted confocal laser endoscope technology to determine the high risk of gastric cancer in real time, instead of tissue biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years undergoing confocal gastroscopy

Exclusion Criteria:

* Patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric disorders who cannot participate in gastroscopy
* Patients with previous surgical procedures on the stomach
* Patients with contraindications to biopsy
* Patients who refuse to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the upper gastrointestinal tract pCLE examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI model in assessing degree of intestinal metaplasia | 2 years
  Pathological biopsy results were used as the gold standard to assess the accuracy of the AI model in diagnosing the degree of intestinal metaplasia at the biopsy site
Sensitivity of AI model to assess degree of intestinal metaplasia | 2 years
  The sensitivity of the AI model to diagnose the degree of intestinal metaplasia at the biopsy site was assessed using pathological biopsy results as the gold standard
Specificity of AI model to assess degree of intestinal metaplasia | 2 years
  Pathological biopsy results were used as the gold standard to assess the specificity of the AI model in diagnosing the degree of intestinal metaplasia at the biopsy site

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China